CLINICAL TRIAL: NCT02504242
Title: A Multi-center, Comparative Clinical Trial to Evaluate the Efficacy and Safety of Inject BMP in Patients Undergoing Transforaminal Lumbar Interbody Fusion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: BioAlpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ExcelOs14-02
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-07

CONDITIONS: Transforaminal Lumbar Interbody Fusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inject BMP (Experimental): ExcelOS Inject / rhBMP-2
  Interventions: Device: Inject BMP
- Locally Harvested Bone (Active Comparator): Locally Harvested Bone
  Interventions: Procedure: Locally Harvested Bone

INTERVENTIONS:
Device: Inject BMP
  Arms: Inject BMP
Procedure: Locally Harvested Bone
  Arms: Locally Harvested Bone

SUMMARY:
A Randomized, Subject-Assessor Blind, Multi-center, Comparative Clinical Trial to evaluate the efficacy and safety of Inject BMP in Patients Undergoing Transforaminal Lumbar Interbody Fusion.

ELIGIBILITY:
Inclusion Criteria:

The subject needs the infusion between the first lumbar vertebrato and the first ilium from those who require posterior spinal instrumentation and interbody fusion for the following reasons,

* Spinal stenosis
* Spinal disc herniation requiring broad laminectomy
* Spondylolisthesis or spondylolysis
* Recurrent herniated disc

Exclusion Criteria:

* Patients with BMD T-score < -3.0
* Women who are pregnant or plan to be pregnant within study period

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Bone Fusion With CT and Dynamic radiographs(X-ray)(post operative 48 weeks) | at 48 weeks after surgery